CLINICAL TRIAL: NCT07007247
Title: Development and Evaluation of a Digital Aftercare Program for Adolescents (12-17 Years) With Depressive Symptoms After Hospital Discharge (Mind-WIN Pilot Study)
Brief Title: Development and Evaluation of a Digital Aftercare Program for Adolescents (12-17 Years) With Depressive Symptoms After Hospital Discharge (Mind-WIN Pilot Study) (Mind-WIN Pilot)
Acronym: MindWinPilot
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Minddistrict GmbH (E-Mental-Health platform) (Unknown); Asklepios Fachklinikum Stadtroda GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mind-Win pilot study; 03DPS1033B (Other Grant/Funding Number: Federal Ministry of Education and Research)
Record Dates: First submitted 2025-05-09; First posted 2025-06-05 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Depressive Disorder; Depression, Unipolar
Keywords: depression; adolescents; aftercare; digital
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mind-Win self-help only (Experimental): Participants are given access to the Mind-WIN aftercare module. The content is completed in self-study including questions for reflection, quiz questions, videos of an experience expert, and audio exercises.
  Interventions: Other: Mind-WIN self-help only
- Mind-Win blended care (Experimental): Participants are given access to the Mind-WIN aftercare module and they get additional therapeutic support (digital contacts). The content of the MIND-WIN aftercare module is completed in self-study including questions for reflection, quiz questions, videos of an experience expert, and audio exercises.
  Interventions: Other: Mind-WIN blended care
- Care-As-Usual (No Intervention): Participants have access to standard medical care through the national health insurance system. After the end of the 18-week comparison period, they also have access to the Mind-WIN self-help module (without therapeutic support).

INTERVENTIONS:
Other: Mind-WIN self-help only — The program lets participants work through the module content at their own speed. Part of the program involves keeping an online diary every two weeks to track symptoms. The results are categorized as mild, moderate, or severe depression. If participants have severe symptoms, the recommendation is to get professional help. If participants are taking medication to improve their depression, they can also use the online diary to track their mood and medication
  Arms: Mind-Win self-help only
Other: Mind-WIN blended care — The program lets participants work through the module content at their own speed. Part of the program involves keeping an online diary every two weeks to track symptoms. The results are categorized as mild, moderate, or severe depression. If participants have severe symptoms, the recommendation is to get professional help. If participants are taking medication to improve their depression, they can also use the online diary to track their mood and medication. In addition to the content provided by the Mind-WIN aftercare module participants get six digital contacts with a psychotherapist.
  Other Names: MindWin blended care
  Arms: Mind-Win blended care

SUMMARY:
Mind-WIN is a digitally supported (app- and web-based) aftercare program for young people between the ages of 12 and 17, which was developed for adolescent patients with depressive symptoms and is intended to be used after inpatient treatment. The aftercare program includes interactive psychoeducational content and exercises on topics such as daily planning, early warning signs, self-care, and goal setting.

This pilot study will assess the feasibility of the study design and methods. It will also examine the preliminary effectiveness of the Mind-WIN aftercare program on self-reported measures compared to the control group. These outcomes include the levels of depressive symptoms, mental health-related quality of life and psychosocial functioning.

Participants are randomly assigned to one of the three study conditions:

1. Mind-WIN self-help only (intervention condition 1): Participants are given access to the Mind-WIN aftercare module. The content is completed in self-study including questions for reflection, quiz questions, videos of an experience expert, and audio exercises.

   .
2. Mind-WIN blended care (intervention condition 2): Participants are given access to the Mind-WIN aftercare module and they get additional therapeutic support (video calls to support the young people during module completion, emotional support and therapeutic conversations).
3. Care-As-Usual (waiting control group): Participants have access to standard medical care through the national health insurance system. At the end of the 18-week comparison period, they also have access to the Mind-WIN aftercare module (without therapeutic support).

Researchers will compare the two Mind-WIN intervention groups (Mind-WIN self-help only and Mind-WIN blended care) to care-as-usual (waiting control group) to answer the following questions:

* Is the study design and methods feasible with the target group?
* Is access to the 12-week Mind-WIN aftercare program associated with greater stabilization in the assessed outcomes (at 12 and 18 weeks) compared to standard care?

ELIGIBILITY:
Inclusion Criteria:

* Recently (maximum four weeks ago) discharged from (partial) inpatient treatment in one of the participating Asklepios clinics
* Age 12 to 17 years
* Main depressive diagnosis:

F32.1 Moderate depressive episode; F32.2 Major depressive episode without psychotic symptoms; F33.1 Recurrent depressive disorder, currently moderate episode; F33.2 Recurrent depressive disorder, currently severe episode without psychotic symptoms

* Ability to give written consent or assent by persons with custody
* Access to a smartphone, tablet or computer with internet access

Exclusion Criteria:

* Mental and behavioural disorders due to psychoactive substance use (ICD-10 codes F10-F19), Schizophrenia, schizotypal and delusional disorders (ICD-10 codes F20-29), major depressive episodes with psychotic symptoms (ICD-10 code F32.3), recurrent depressive disorder, current severe episode with psychotic symptoms (ICD-10 code F33.3)
* acute suicidality
* bipolar disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
depressive symptoms (PHQ-A) at 12 weeks | 12 weeks after baseline
  Note: As this is a pilot study, no separation into primary and secondary outcomes are formulated at this stage. We define the current primary outcome due to system requirements.
  PHQ-A total score:
  0-4 (minimal depression) 5-9 (mild depression) 10-14 (moderate depression) 15-19 (moderately severe depression) 20-27 (severe depression)

SECONDARY OUTCOMES:
anxiety and depressive symptoms (RCADS-25) at 12 weeks | 12 weeks after baseline
  Revised Children's Anxiety and Depression Scale (RCADS-25) total depression and anxiety score (range 0 to 75, higher scores represent more symptoms)
anxiety symptoms (GAD-7) at 12 weeks | 12 weeks after baseline
  GAD-7 total score:
  0-4 (minimal anxiety) 5-9 (mild anxiety) 10-14 (moderate anxiety) 15-21 (severe anxiety)
mental health-related quality of life (KIDSCREEN-10) at 12 weeks | 12 weeks after baseline
  global Health-Related Quality-of-Life (HRQoL) index (T-values)
psychosocial functioning (SDQ - self-completion) at 12 weeks | 12 weeks after baseline
  total difficulties score (range 0 to 40, higher scores represent more difficulties)
Avoiding school/training at 12 weeks | 12 weeks after baseline
  number of days absent since baseline
medication adherence at 12 weeks | 12 weeks after baseline
  report if medication was taken as prescribed (yes or no response)
transfer knowledge from psychiatry treatment baseline at 12 weeks | 12 weeks after baseline
  level of transfer knowledge from psychiatry since baseline (score between 0 and 4, higher score represents higher transfer)
inpatient treatment psychiatry at 12 weeks | 12 weeks after baseline
  report of inpatient treatment in a psychiatric hospital since baseline (yes or no response)
ZUF-8 at 12 weeks (only Intervention groups) | 12 weeks after baseline
  total score ZUF-8 (indicating patients satisfaction): high scale values indicate high "satisfaction", low scale values indicate low "satisfaction".
depressive symptoms (PHQ-A) at 18 weeks | 18 weeks after baseline
  PHQ-A total score:
  0-4 (minimal depression) 5-9 (mild depression) 10-14 (moderate depression) 15-19 (moderately severe depression) 20-27 (severe depression)
anxiety and depressive symptoms (RCADS-25) at 18 weeks | 18 weeks after baseline
  RCADS-25 total depression and anxiety score (range 0 to 75, higher scores represent more symptoms)
anxiety symptoms (GAD-7) at 18 weeks | 18 weeks after baseline
  GAD-7 total score:
  0-4 (minimal anxiety) 5-9 (mild anxiety) 10-14 (moderate anxiety) 15-21 (severe anxiety)
mental health-related quality of life (KIDSCREEN-10) at 18 weeks | 18 weeks after baseline
  global HRQoL index (T-values)
psychosocial functioning (SDQ - self-completion) at 18 weeks | 18 weeks after baseline
  total difficulties score (range 0 to 40, higher scores represent more difficulties)
avoiding school/training at 18 weeks | 18 weeks after baseline
  number of days absent since baseline
medication adherence at 18 weeks | 18 weeks after baseline
  report if medication was taken as prescribed (yes or no response)
transfer knowledge frompsychiatry treatment baseline at 18 weeks | 18 weeks after baseline
  level of transfer knowledge from psychaitry since baseline (score between 0 and 4, higher score represents higher transfer)
inpatient treatment psychiatry at 18 weeks | 18 weeks after baseline
  report of inpatient treatment in a psychiatry hospital since baseline (yes or no response)

CONTACTS AND LOCATIONS:
Overall Officials: Holger Schulz, Prof., Study Director — Universitätsklinikum Hamburg-Eppendorf; Martin Schumm, Dr., Principal Investigator — Asklepios Clinic Stadtroda
Locations (3):
- Germany (3):
  - Asklepios Klinikum Harburg, Hamburg
  - Asklepios Fachklinikum Lübben, Lubin
  - Asklepios Fachklinikum Stadtroda, Stadtroda

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to data protection laws.